CLINICAL TRIAL: NCT02905630
Title: Effect of Aerobic High-intensity Exercise Training on Coronary Flow Reserve and Endothelial Function in Individuals With Chest Pain and Normal Coronary Angiogram
Brief Title: The Syndrome X-ercise Study SYNDEX
Acronym: SYNDEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: University of Bergen (Other); University of Stavanger (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 362Syndex
Record Dates: First submitted 2016-08-24; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Angina
Keywords: coronary flow reserve; angina; exercise training
MeSH Terms: conditions — Angina Pectoris | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): High intensity aerobic exercise training
  Interventions: Other: Exercise training
- No training (No Intervention): No exercise training, only ordinary daily life activities.

INTERVENTIONS:
Other: Exercise training — high intensity aerobic interval training
  Arms: Exercise training

SUMMARY:
This pilot study evaluates the effect of exercise training on CFR, functional capacity, heart rate variability, endothelial function and quality of life in patients with no obstructive coronary artery disease and angina.

DETAILED DESCRIPTION:
Impaired coronary flow reserve (CFR) is associated with increased mortality in patients with chest pain despite normal coronary arteries (chest pain and normal coronary angiograms (CPNCA)) , . Furthermore, impaired CFR without any concomitant impairment of regional or global left ventricular function have additional prognostic significance . In patients with hypertension both microvascular dysfunction and increased left ventricular mass (LVM) are described sequels . LVM has also been associated with endothelial dysfunction and coronary artery remodelling . In addition, patients with hypertrophic obstructive cardiomyopathy (HOCM) and an impaired micro vascular cardiac circulation assessed with PET, have been documented to have a poor prognosis . Also diastolic dysfunction as measured by Em/Am ratio during stress dobutamine echocardiography is related to CFR . Patients with Diabetes Mellitus have an impaired prognosis and longstanding disease influence microvascular physiology . Several methods have been utilized to assess micro vascular function including intracoronary Doppler measurements. CRF can now be assessed with transthoracic Doppler registration .

Several patients with angina and normal coronary arteries show persistence and even worsening of angina symptoms over time. . These patients constitute a therapeutic problem with considerable residual morbidity associated with functional limitation and reduced quality of life . The primary end point in the treatment of these patients is symptom control .

Reduced physical activity is one of the major avoidance behaviours in patients with coronary heart disease . On the other hand several studies have documented the positive effect of ET in this population . Psychological morbidity with great impact on daily living is well known in both patients with cardiovascular disease and in patients with chest pain with no obvious physical disease. This includes patients with CPNCA. These patients constitute a relatively large proportion of patients taken care of by the health authority system indicating that this issue has economic consequences for the society that is not neglectable2.

Exercise training (ET) has been shown to improve endothelial function in patients with coronary artery disease (CAD) and to reduce LVM in hypertension.. ET also improves endothelial dysfunction and reverse inflammation in CAD. It is also associated with improved outcome in the general population and in patients with CAD and heart failure. It has been documented that hs-CRP correlates with symptoms and ECG markers of myocardial ischemia in CPNCA patients . Whether hs-CRP is related to the pathogenesis of angina in these patients deserves further investigation. Whether ET may influence on pathological reduced CFR is currently not known.

Interventions proposed in CPNCA patients are directed at either improving microvascular function or decreasing chest pain perception, in an attempt to counteract the accepted pathophysiological mechanisms of the syndrome. A multidisciplinary approach and a genuine, sympathetic appreciation by the health staff of the devastating effect of cardiac syndrome X on the patients' quality of life usually have a positive therapeutic impact . Unfortunately, most treatments have been evaluated in small numbers of patients and/or in uncontrolled trials, thus making it difficult to establish their real degree of effectiveness. Tynni Lee 11 investigated the effects of physical training and relaxation therapy on exercise capacity and quality of life in patients with syndrome X. It is the first trial reported to assess the effect of physiotherapy intervention in terms of quality of life in patients with coronary syndrome X. Female patients with this syndrome benefit from physical training in terms of exercise capacity and quality of life, and from relaxation therapy in terms of quality of life. However a limitation is the small sample size and therefore non-significant findings may be due to an inability to detect a difference among groups. Further studies with larger number of patients are recommended. Different modes of physiotherapy could have the potential to break the vicious circle of effort-induced chest pain, functional limitations and poor quality of life in the patients with coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* outpatients and patients admitted to the hospital with a history of repeated episodes of exercise induced chest pain.
* normal or near normal coronary angiogram or negative CT coronary angiogram
* age > 18 years
* being able to participate in training groups 3 times a week.

Exclusion Criteria:- Prior myocardial infarction

* serious valve disease
* cancer
* previous radiation or drug therapy for cancer
* musculoskeletal problems making ET impossible
* ongoing serious inflammatory disease
* intracardiac devices
* presumed insufficient acoustic windows because of severe emphysema or gross overweight
* atrial fibrillation
* participation in other ongoing studies.
* contrast allergy
* contraindication to adenosine infusion
* vasospasm angina

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve | 3 months
  Changes of Cornary flow reserve following 3 months of exercise training

SECONDARY OUTCOMES:
Endothelial function | 3 months
  Arterial diameter after occlusion at baseline and at 3 months follow up
Functional capacity | 3 months
  Changes in cardiopulmonary exercise testing following 3 months of exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Alf Inge Larsen, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen AI, Saeland C, Vegsundvag J, Skadberg MS, Nilsen J, Butt N, Ushakova A, Valborgland T, Munk PS, Isaksen K. Aerobic high-intensity interval exercise training in patients with angina and no obstructive coronary artery disease: feasibility and physiological effects. Eur Heart J Open. 2023 Mar 22;3(2):oead030. doi: 10.1093/ehjopen/oead030. eCollection 2023 Mar. PMID 37113515